CLINICAL TRIAL: NCT02220998
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Compare the Efficacy and Safety of Sofosbuvir/GS-5816 Fixed Dose Combination for 12 Weeks With Sofosbuvir and Ribavirin for 12 Weeks in Subjects With Chronic Genotype 2 HCV Infection
Brief Title: Comparison of Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks With Sofosbuvir and Ribavirin for 12 Weeks in Adults With Chronic Genotype 2 HCV Infection
Acronym: ASTRAL-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1139
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2016-09

CONDITIONS: Hepatitis C Virus Infection
Keywords: Hepatitis C; HCV; cirrhosis; Sofosbuvir; Sovaldi; SOF/VEL; GS-5816; GS-7977; liver; Treatment naive; Treatment Experience; genotype 2
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — sofosbuvir-velpatasvir drug combination; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOF/VEL (Experimental): SOF/VEL FDC for 12 weeks
  Interventions: Drug: SOF/VEL
- SOF+RBV (Experimental): SOF+RBV for 12 weeks
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL — SOF/VEL (400/100 mg) FDC tablet administered orally once daily
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: SOF/VEL
Drug: SOF — SOF 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: SOF+RBV
Drug: RBV — RBV tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: SOF+RBV

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) for 12 weeks compared to treatment with sofosbuvir (SOF) plus ribavirin (RBV) for 12 weeks in participants with chronic genotype 2 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL
* HCV genotype 2
* Chronic HCV infection (≥ 6 months)
* Females of childbearing potential must have a negative serum pregnancy test
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Must be of generally good health, with the exception of chronic HCV infection, as determined by the investigator.

Exclusion Criteria:

* Current or prior history of clinically-significant illness (other than HCV that may interfere with treatment, assessment or compliance with the protocol;
* Screening electrocardiogram (ECG) with clinically significant abnormalities
* Laboratory results outside of acceptable ranges at Screening
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency, cholangitis)
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anu Osinusi, MD, Study Director — Gilead Sciences
Locations (40):
- United States (39):
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Pasadena, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Bradenton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Emory university, Atlanta, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Monroe, Louisiana
  - Baltimore, Maryland
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Santa Fe, New Mexico
  - Great Neck, New York
  - New York, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Asselah T, Charlton M, Feld J, Foster GR, Mcnally J, Brainard DM, et al. The ASTRAL Studies: Evaluation of SOF/GS-5816 Single Tablet Regimen for the Treatment of Genotype 1-6 HCV Infection [Poster P1332]. J Hepatol 2015;62:S855-S6.
- [Result] Sulkowski, MS., Brau N., Lawitz E., Shiffman ML, Towner WL, Ruane PJ et al. A Randomized Controlled Trial of Sofosbuvir/GS-5816 Fixed Dose Combination for 12 Weeks Compared to Sofosbuvir with Ribavirin for 12 Weeks in Genotype 2 HCV Infected Patients: The Phase 3 ASTRAL-2 Study [Oral 205] Hepatology 2015; 62: 1 (SUPPL) 313A.
- [Result] Foster GR, Afdhal N, Roberts SK, Brau N, Gane EJ, Pianko S, Lawitz E, Thompson A, Shiffman ML, Cooper C, Towner WJ, Conway B, Ruane P, Bourliere M, Asselah T, Berg T, Zeuzem S, Rosenberg W, Agarwal K, Stedman CA, Mo H, Dvory-Sobol H, Han L, Wang J, McNally J, Osinusi A, Brainard DM, McHutchison JG, Mazzotta F, Tran TT, Gordon SC, Patel K, Reau N, Mangia A, Sulkowski M; ASTRAL-2 Investigators; ASTRAL-3 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 2 and 3 Infection. N Engl J Med. 2015 Dec 31;373(27):2608-17. doi: 10.1056/NEJMoa1512612. Epub 2015 Nov 17. PMID 26575258
- [Derived] Jacobson IM, Bourgeois S, Mathurin P, Thuluvath P, Ryder SD, Gerken G, Hernandez C, Vanstraelen K, Scherbakovsky S, Osinusi A, Tedesco D, Foster GR. The tolerability of sofosbuvir/velpatasvir for 12 weeks in patients treated in the ASTRAL 1, 2 and 3 studies: A pooled safety analysis. J Viral Hepat. 2023 May;30(5):448-454. doi: 10.1111/jvh.13814. Epub 2023 Mar 2. PMID 36740893
- [Derived] Younossi ZM, Stepanova M, Feld J, Zeuzem S, Sulkowski M, Foster GR, Mangia A, Charlton M, O'Leary JG, Curry MP, Nader F, Henry L, Hunt S. Sofosbuvir and Velpatasvir Combination Improves Patient-reported Outcomes for Patients With HCV Infection, Without or With Compensated or Decompensated Cirrhosis. Clin Gastroenterol Hepatol. 2017 Mar;15(3):421-430.e6. doi: 10.1016/j.cgh.2016.10.037. Epub 2016 Nov 12. PMID 27847279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 22 September 2014. The last study visit occurred on 03 September 2015.
Pre-assignment Details: 317 participants were screened.
Groups:
- SOF/VEL: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet administered orally once daily for 12 weeks
- SOF+RBV: Sofosbuvir (SOF) 400 mg tablet administered orally once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL | SOF+RBV
Started | 135 | 134
Completed | 128 | 123
Not Completed | 7 | 11
Not completed — Randomized but Never Treated | 1 | 2
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 0 | 5
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug.
Groups:
- SOF/VEL: SOF/VEL (400/100 mg) FDC tablet administered orally once daily for 12 weeks
- SOF+RBV: SOF 400 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL | SOF+RBV | Total
Number analyzed (Participants) | 134 | 132 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10.6) | 57 (9.3) | 57 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 60 | 108
  Male | 86 | 72 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 23 | 49
  Not Hispanic or Latino | 104 | 107 | 211
  Unknown or Not Reported | 4 | 2 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 6 | 12 | 18
  White | 124 | 111 | 235
  Asian | 1 | 5 | 6
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Other | 1 | 2 | 3
  Not Disclosed | 2 | 1 | 3
Cirrhosis Status [Number; unit: participants]
  Present | 19 | 19 | 38
  Absent | 115 | 112 | 227
  Missing | 0 | 1 | 1
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 55 | 46 | 101
    CT | 61 | 64 | 125
    TT | 18 | 22 | 40
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.78) | 6.4 (0.74) | 6.4 (0.76)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 23 | 31 | 54
  ≥ 800,000 IU/mL | 111 | 101 | 212

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants randomized or enrolled into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF+RBV
Number analyzed (Participants) | 134 | 132
percentage of participants | 99.3 [95.9 to 100.0] | 93.9 [88.4 to 97.3]
Statistical Analysis 1: Comparison: SOF/VEL vs SOF+RBV; Test type: Non-Inferiority or Equivalence — A sample size of 120 per treatment group provided 90% power to establish non-inferiority in the SVR12 rates between the SOF/VEL group and the SOF+RBV group. It was based on the assumptions that the non-inferiority margin is 10%, both groups have a SVR12 rate of 94%, and the significance level is 0.025 one-sided; Difference in proportions = 5.2, 95% CI 2-sided [0.2 to 10.3] — Difference in proportions between treatment groups and associated 95% confidence intervals (CI) are calculated based on stratum-adjusted Mantel-Haenszel proportions
Statistical Analysis 2: Comparison: SOF/VEL vs SOF+RBV; The superiority of SOF/VEL for 12 weeks over SOF+RBV for 12 weeks was to be tested if the efficacy of SOF/VEL for 12 weeks was demonstrated to be statistically noninferior to SOF+RBV for 12 weeks (ie, if the lower bound of the 95% CI for the strata-adjusted difference in the proportions between groups was greater than the prespecified noninferiority margin of -10%); Test type: Superiority or Other; p = 0.018, Cochran-Mantel-Haenszel — P-value was stratified by cirrhosis status and prior treatment experience

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | SOF+RBV
Number analyzed (Participants) | 134 | 132
percentage of participants | 0.7 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF+RBV
Number analyzed (Participants) | 134 | 132
percentage of participants
  SVR4 | 99.3 [95.9 to 100.0] | 96.2 [91.4 to 98.8]
  SVR24 | 99.3 [95.9 to 100.0] | 93.9 [88.4 to 97.3]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 6, 8, 10, and 12
Time Frame: Weeks 1, 2, 4, 6, 8, 10, and 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF+RBV
Number analyzed (Participants) | 134 | 132
percentage of participants
  Week 1 (SOF/VEL: N = 133; SOF+RBV: N = 132) | 12.8 [7.6 to 19.7] | 22.7 [15.9 to 30.8]
  Week 2 (SOF/VEL: N = 133; SOF+RBV: N = 132) | 57.1 [48.3 to 65.7] | 59.8 [51.0 to 68.3]
  Week 4 (SOF/VEL: N = 133; SOF+RBV: N = 132) | 90.2 [83.9 to 94.7] | 90.2 [83.7 to 94.7]
  Week 6 (SOF/VEL: N = 133; SOF+RBV: N = 132) | 97.7 [93.5 to 99.5] | 99.2 [95.9 to 100.0]
  Week 8 (SOF/VEL: N = 133; SOF+RBV: N = 132) | 100.0 [97.3 to 100.0] | 100.0 [97.2 to 100.0]
  Week 10 (SOF/VEL: N = 133; SOF+RBV: N = 132) | 100.0 [97.3 to 100.0] | 100.0 [97.2 to 100.0]
  Week 12 (SOF/VEL: N = 133; SOF+RBV: N = 131) | 100.0 [97.3 to 100.0] | 100.0 [97.2 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 6, 8, 10, and 12
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 10, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF+RBV
Number analyzed (Participants) | 134 | 132
log10 IU/mL
  Change at Wk 1 (SOF/VEL: N= 132; SOF+RBV: N= 131) | -4.51 (0.666) | -4.51 (0.553)
  Change at Wk 2 (SOF/VEL: N= 132; SOF+RBV: N= 131) | -5.08 (0.761) | -5.04 (0.701)
  Change at Wk 4 (SOF/VEL: N= 132; SOF+RBV: N= 131) | -5.29 (0.781) | -5.24 (0.755)
  Change at Wk 6 (SOF/VEL: N= 133; SOF+RBV: N= 131) | -5.31 (0.781) | -5.27 (0.741)
  Change at Wk 8 (SOF/VEL: N= 133; SOF+RBV: N= 132) | -5.32 (0.782) | -5.27 (0.739)
  Change at Wk 10 (SOF/VEL: N= 133; SOF+RBV: N= 132) | -5.32 (0.782) | -5.27 (0.739)
  Change at Wk 12 (SOF/VEL: N= 133; SOF+RBV: N= 131) | -5.32 (0.782) | -5.26 (0.737)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | SOF+RBV
Number analyzed (Participants) | 134 | 132
percentage of participants | 0 | 4.5

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL | SOF+RBV
Serious Adverse Events (participants affected / at risk) | 2/134 | 2/132
Other Adverse Events (participants affected / at risk) | 69/134 | 84/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=134) | SOF+RBV (N=132)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=134) | SOF+RBV (N=132)
Anaemia (Blood and lymphatic system disorders) | 0 | 8
Abdominal pain (Gastrointestinal disorders) | 5 | 7
Nausea (Gastrointestinal disorders) | 14 | 20
Vomiting (Gastrointestinal disorders) | 5 | 8
Fatigue (General disorders) | 20 | 47
Nasopharyngitis (Infections and infestations) | 8 | 2
Sinusitis (Infections and infestations) | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 8 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Dizziness (Nervous system disorders) | 3 | 8
Headache (Nervous system disorders) | 24 | 29
Anxiety (Psychiatric disorders) | 8 | 8
Insomnia (Psychiatric disorders) | 6 | 19
Irritability (Psychiatric disorders) | 4 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 7
Rash (Skin and subcutaneous tissue disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years